CLINICAL TRIAL: NCT00707512
Title: INFORM: Investigating Natalizumab Through Further Observational Research and Monitoring
Brief Title: CD INFORM: Investigating Natalizumab Through Further Observational Research and Monitoring
Acronym: INFORM
Status: Terminated | Type: Observational
Why Stopped: Sponsor's decision.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 101CD401; ELN100226-CD451 (Other: Elan Pharmaceuticals)
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: natalizumab — Administered as specified in the TOUCH Prescribing Program
  Other Names: Tysabri; BG00002

SUMMARY:
The primary objective of the study is to determine the incidence and pattern of serious and/or clinically significant infections, malignancies, and other serious adverse event (SAE) in participants with Crohn's Disease (CD) treated with natalizumab. The secondary objective of this study in this study population is to evaluate disease severity over time in participants with CD treated with natalizumab based on changes in the Harvey-Bradshaw Index (HBI).

DETAILED DESCRIPTION:
This study was originally conducted by Elan Pharmaceuticals, Inc. (Elan) in collaboration with Biogen under a protocol written by Elan. Biogen is solely responsible for the study since April 2013.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with Crohn's Disease (CD) who are eligible for therapy according to US Tysabri label and who are enrolled in the Tysabri Outreach Unified Commitment to Health (TOUCH) Prescribing Program.

Key Exclusion criteria:

* None

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CD who were naïve to natalizumab treatment and participants with CD who have been previously treated with natalizumab.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2008-06-30 (Actual); Primary Completion 2015-05-28 (Actual); Study Completion 2015-05-28 (Actual)

PRIMARY OUTCOMES:
Rate of serious and/or clinically significant infections, malignancies, and other SAEs in participants with Crohn's Disease treated with natalizumab | Every 6 months for up to 5 years following the first Tysabri infusion

SECONDARY OUTCOMES:
Measurement of disease severity over time as assessed by change in HBI | Every 6 months for up to 5 years following the first Tysabri infusion

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (35):
- United States (34):
  - Research site, Scottsdale, Arizona
  - Research site, Oceanside, California
  - Research site, San Francisco, California
  - Research site, Hamden, Connecticut
  - Research site, Hartford, Connecticut
  - Research site, Gainesville, Florida
  - Research site, Miami, Florida
  - Research site, Winter Park, Florida
  - Research site, Atlanta, Georgia
  - Research site, Crestview Hills, Kentucky
  - Research site, Lexington, Kentucky
  - Research site, Louisville, Kentucky
  - Research site, Baltimore, Maryland
  - Research site, Boston, Massachusetts
  - Research site, Ann Arbor, Michigan
  - Research site, Plymouth, Minnesota
  - Research site, Columbia, Missouri
  - Research site, Lebanon, New Hampshire
  - Research site, Egg Harbor, New Jersey
  - Research site, Great Neck, New York
  - Research site, Lake Success, New York
  - Research site, New York, New York
  - Research site, Rochester, New York
  - Research site, Troy, New York
  - Research site, Chapel Hill, North Carolina
  - Research site, Charlotte, North Carolina
  - Research site, Raleigh, North Carolina
  - Research site, Cincinnati, Ohio
  - Research site, Cleveland, Ohio
  - Research site, Providence, Rhode Island
  - Research site, Nashville, Tennessee
  - Research site, Grapevine, Texas
  - Research site, Houston, Texas
  - Research site, Tacoma, Washington
- Research site, San Juan, Puerto Rico